CLINICAL TRIAL: NCT03810638
Title: Creation of a Digital Heart Failure Registry Using a Novel Mobile Health Platform: HUGO-HF
Acronym: HUGO-HF
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 2000024317
Record Dates: First submitted 2019-01-17; First posted 2019-01-22 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-08

CONDITIONS: Heart Failure
Keywords: Heart Failure; Heart Transplant; Left Ventricular Assist Device
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Heart Failure Patients: All Heart Failure Patients seen at 3 major academic medical centers.

SUMMARY:
The investigators goal is to create a digital registry that allows for seamless integration of patient reported outcomes, electronic health record data, and pharmacy information into data collection. The investigators will accomplish this using a novel patient centered mobile health platform called Hugo that will allow them to engage patients in an entirely novel manner.

DETAILED DESCRIPTION:
Heart failure is the most common cause of mortality and morbidity in the United States and in Western Europe. It is a complex and chronic illness, and patient journeys vary considerably. However, to date, guidance about how to best treat patients has relied on large clinical international trials that do not represent contemporary patients and only include snapshots of the syndrome-at times when the patients interact with the health care system. Additionally, patient participation in clinical research in the US is extremely low, approximated at 3% in cancer and far lower for disease states such as heart failure.

One of the key reasons for this is a lack of patient engagement and trust in the research enterprise, especially among the elderly and minorities, groups that are disproportionally impacted by heart failure. To address this, the investigators plan to test a novel patient-powered, smartphone-based mobile health platform (called Hugo) developed at Yale School of Medicine for real-world surveillance of patient reported outcomes in heart failure patients treated at 3 Major Academic Medical Centers. Participants will then be queried about specific symptoms and health conditions at enrollment and prespecified time points for 2 years. The subgroup of participants who own devices that track their activity data will have the option of syncing them to this mobile health platform to provide additional insights into their health and health outcomes. Additionally, participants will have the option to learn about opportunities to participate in heart failure clinical research. This digital registry will also allow seamless integration of patient reported outcomes, electronic health record (EHR) data, and pharmacy information into data collection.

Overall, the aim for this study is to create a digital registry using a novel patient centered mobile health platform of heart failure patients across large health care systems that allows investigators to engage patients in an entirely novel manner.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 Years
* English Speaking
* Diagnosis of heart failure
* Participant is willing and able to read and sign consent and participate in study
* Participant has an email account

Exclusion Criteria:

- Unable to participate in registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will aim to recruit patients who are admitted to the hospital with a diagnosis of heart failure at or seen in the heart failure clinic.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in Quality of Life using the KCCQ-12 | 2 Years
  Short Version of the KCCQ will be used. The Kansas City Cardiomyopathy Questionnaire (KCCQ) is the most validated instrument to measure quality of life in heart failure.

SECONDARY OUTCOMES:
Hospitalizations | 2 years
  All-cause hospitalizations among patients in registry
Death | 2 years
  Rates of death among patients in registry
Medication Usage | 2 years
  Use of guideline directed medical therapies will be done by automatically syncing the patients portal with pharmacy data to provide the most uptodate medication information.
Activity Details | 2 years
  Activity information based on synced devices

CONTACTS AND LOCATIONS:
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahmad T, Freeman JV, Asselbergs FW. Can advanced analytics fix modern medicine's problem of uncertainty, imprecision, and inaccuracy? Eur J Heart Fail. 2019 Jan;21(1):86-89. doi: 10.1002/ejhf.1370. Epub 2018 Dec 10. No abstract available. PMID 30537243
- [Result] Krumholz HM. Big data and new knowledge in medicine: the thinking, training, and tools needed for a learning health system. Health Aff (Millwood). 2014 Jul;33(7):1163-70. doi: 10.1377/hlthaff.2014.0053. PMID 25006142
- [Result] Bhavnani SP, Parakh K, Atreja A, Druz R, Graham GN, Hayek SS, Krumholz HM, Maddox TM, Majmudar MD, Rumsfeld JS, Shah BR. 2017 Roadmap for Innovation-ACC Health Policy Statement on Healthcare Transformation in the Era of Digital Health, Big Data, and Precision Health: A Report of the American College of Cardiology Task Force on Health Policy Statements and Systems of Care. J Am Coll Cardiol. 2017 Nov 28;70(21):2696-2718. doi: 10.1016/j.jacc.2017.10.018. No abstract available. PMID 29169478
- See also: A Novel Digital Platform for Research — http://hugophr.com/